CLINICAL TRIAL: NCT00012922
Title: Low Literacy Intervention for Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: PCI 99-158
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Low Literacy Intervention for Colorectal Cancer Screening

INTERVENTIONS:
Behavioral: Low Literacy Intervention for Colorectal Cancer Screening

SUMMARY:
Of 17 performance measures of hospital quality regularly reported for the Veterans Administration (VA) health care system, rates of colorectal cancer screening are the lowest.

DETAILED DESCRIPTION:
Background:

Of 17 performance measures of hospital quality regularly reported for the Veterans Administration (VA) health care system, rates of colorectal cancer screening are the lowest.

Objectives:

The objectives of this study were to 1) test whether a health care provider-directed intervention increased colorectal cancer screening rates in an urban VA medical center and 2) evaluate the cost-effectiveness of the intervention.

Methods:

The study was a randomized controlled trial, conducted at two clinic firms at a VA Medical Center in Chicago. Eligible patients were men, age 50 and older, had no personal or family history of colorectal cancer or polyps, had not received colorectal cancer screening, and had at least one visit to the clinic during the study period. Health care providers in the intervention firm attended a workshop on colorectal cancer screening. Every 4-6 months they attended quality improvement workshops where they received group screening rates, individualized confidential feedback, and training on improving communication with patients with limited literacy skills. Medical records were reviewed for colorectal cancer screening recommendations and completion. Literacy level was assessed in a subset of patients. In the cost-effectiveness analysis, resource and cost estimates were derived.

Status:

The project is complete.

ELIGIBILITY:
Inclusion Criteria:

Patients over 50 with average risk for colorectal cancer. Patients with family history and/or personal history excluded, as well as those up to date on colorectal cancer screening.

Exclusion Criteria:

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Bennett, MD PhD MPP, Principal Investigator — Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL, Chicago, Illinois, United States